CLINICAL TRIAL: NCT01872819
Title: Treatment for Relapsed/Refractory AML Based on a High Throughput Drug Sensitivity Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pamela S Becker, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8003; NCI-2013-01070 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 8003 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Chronic Myelomonocytic Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Refractory Anemia With Excess Blasts
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Myelomonocytic, Chronic; Myeloproliferative Disorders; Anemia, Refractory, with Excess of Blasts | interventions — Drug Screening Assays, Antitumor; Drug Therapy; Biological Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy, biological therapy) (Experimental): Patients receive 1 of 160 possible interventions based on high throughput drug sensitivity assay.
  Interventions: Other: antitumor drug screening assay; Drug: chemotherapy; Biological: biological therapy

INTERVENTIONS:
Other: antitumor drug screening assay — Undergo high throughput drug sensitivity assay
  Other Names: antitumor drug screening assays; drug screening assays, antitumor
Drug: chemotherapy — Patients receive 1 of 160 possible interventions
  Other Names: chemo
Biological: biological therapy — Patients receive 1 of 160 possible interventions

SUMMARY:
This clinical trial uses a laboratory test called a high throughput sensitivity assay in planning treatment for patients with relapsed or refractory acute myeloid leukemia. The aim is to try to identify drugs that may be effective in killing leukemia cells for those patients who will not be cured with conventional chemotherapy. This assay will test multiple drugs simultaneously against a patient's own donated blood sample. The goal is to use this laboratory assay to best match a drug to a patient's disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain results from a high throughput drug sensitivity assay within 10 days, procure drug within 14 days and initiate treatment within 21 days.

SECONDARY OBJECTIVES:

I. To achieve a response (cytoreduction or at least partial response) greater that than expected for comparable refractory patient populations with other salvage regimens.

OUTLINE:

A patient receives a drug intervention based on the results of a high throughput sensitivity assay. This assay best matches a drug to the patient's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia by World Health Organization (WHO) criteria (except acute promyelocytic leukemia), acute leukemias of ambiguous lineage by WHO criteria, or myelodysplastic syndrome refractory anemia with excess blasts (RAEB)-2 by WHO classification or advanced myeloproliferative neoplasm with >= 10% blasts in the bone marrow or peripheral blood, including chronic myelomonocytic leukemia (CMML)-2 by WHO classification who have failed 2 inductions at initial diagnosis or failed >= 2 salvage regimens for relapsed acute myeloid leukemia (AML)
* Patients who have had a 1st remission for >= 1 year must have received cytotoxic chemotherapy as a salvage regimen
* Eastern Cooperative Oncology Group (ECOG) performance status 0 - 3
* Expectation that we can obtain about 100 million blasts from blood and/or marrow (for example, circulating blast count of 5,000 or greater)
* Bilirubin =< 1.5 x institutional upper limit of normal (IULN) unless elevation is thought to be due to Gilbert's syndrome, hemolysis, or hepatic infiltration by the hematologic malignancy
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) and serum pyruvate glutamate transaminase (SPGT) (alanine aminotransferase [ALT]) =< 2.5 x IULN, unless elevation in thought to be due to hepatic infiltration by the hematologic malignancy
* Alkaline phosphatase =< 2.5 X ULN
* Serum creatinine =< 2.0 mg/dL
* Stable or improving on appropriate antimicrobial therapy for infection, without ongoing fever
* Informed consent
* Willing to use contraception

Exclusion Criteria:

* No other concomitant treatment for leukemia
* No other active cancer that requires systemic chemotherapy or radiation
* Significant organ compromise that will increase risk of toxicity or mortality
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-08-02 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-11-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Becker, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy, Biological Therapy): Patients receive 1 of 160 possible interventions based on high throughput drug sensitivity assay.
  antitumor drug screening assay: Undergo high throughput drug sensitivity assay
  chemotherapy: Patients receive 1 of 160 possible interventions
  biological therapy: Patients receive 1 of 160 possible interventions
  16 patients were enrolled. 14 patients were treated.
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Biological Therapy)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: relapsed, refractory AML patients. 16 patients were enrolled, 14 patients were treated.
Arm/Group | Treatment (Chemotherapy, Biological Therapy)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Achievability of Performing Individualized Drug Screening and Initiating Therapy Based on the Results of the Drug Screen for Poor Risk Patients With Relapsed or Refractory AML
Description: Whether treatment was administered in the time frame based on the high throughput drug screen. Time from sample procurement to assay results.
Time Frame: Up to 21 days
Population: 14 patients were treated.
Measure: Median (Full Range); unit: days
Groups:
- Treated Patients: 14 patients were treated.
Arm/Group | Treated Patients
Number analyzed (Participants) | 14
days | 5.1 [4 to 8]

2. Secondary Outcome: Rate of Complete Response, Defined by Criteria of Cheson et al.
Description: Number of patients who achieved a Complete Response (CR) with Minimal Residual Disease (MRD), a Complete Response with incomplete hematologic recovery (CRi), or showed reduced blasts in their bone marrow by flow cytometry (Cytoreduction).
  Cheson et al. defines a CR as: Bone Marrow blasts <5%, absence of circulating blasts and blasts with Auer rods, absence of extramedullary disease, absolute neutrophil count >1.0 x 10^9/L, and platelet count >100 x 10^9/L. Cheson et al. defines a CRi as: all CR criteria except for residual neutropenia (<1.0 x 10^9/L) or thrombocytopenia (<100 x 10^9/L).
Time Frame: Baseline up to 2 years
Population: 14 patients received therapy. Out of 14 patients treated, 9 were evaluable (4 patients died prior to D14-21 marrow and 1 patient refused the D14-21 marrow).
Measure: Number; unit: Patients
Arm/Group | Treated Patients
Number analyzed (Participants) | 9
Patients
  CR with MRD | 1
  CRi | 2
  Cytoreduction | 6

ADVERSE EVENTS:
Time Frame: 2 years
Description: Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Treatment (Chemotherapy, Biological Therapy)
Serious Adverse Events (participants affected / at risk) | 11/14
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Biological Therapy) (N=14)
seizure (Nervous system disorders) | 2 (2) — due to thrombocytopenia due to underlying disease
pneumonia (Infections and infestations) | 1 (1) — fungal
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1) — secondary to blast crisis
malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
febrile neutropenia (Infections and infestations) | 5 (7)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
hypokalemia (Investigations) | 2 (2) — intermittent
confusion (Psychiatric disorders) | 1 (1) — intermittent
hyperbilirubinemia (Investigations) | 2 (2)
Hypoalbuminemia (Investigations) | 1 (1)
pneumonia (Infections and infestations) | 1 (1) — stenotrophomonas maltophilia
febrile neutropenia (Infections and infestations) | 1 (1) — intermittent
drug rash (Skin and subcutaneous tissue disorders) | 1 (1)
hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) — intermittent
mucositis (Gastrointestinal disorders) | 1 (2)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
blood bilirubin increased (Investigations) | 1 (1)
bacteremia-GPC (Infections and infestations) | 1 (1)
sepsis (Infections and infestations) | 1 (1) — Neutropenic secondary to GNR bacteremia
hypotension (Vascular disorders) | 2 (2)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) — intermittent
tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2)
pleural effusions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
worsening abdominal pain (Gastrointestinal disorders) | 1 (1)
severe bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
c-diff colitis infection (Infections and infestations) | 1 (1)
LE edema (General disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — related to pleural effusion
coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Elevated AST (Investigations) | 1 (1)
DIC (Blood and lymphatic system disorders) | 1 (1)
uric acid (Metabolism and nutrition disorders) | 1 (1)
acute systolic heart failure (Cardiac disorders) | 1 (1)
cardiogenic shock (Cardiac disorders) | 1 (1)
hypoxemic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
refractory hypotension (Vascular disorders) | 1 (1)
refractory shock (General disorders) | 1 (1)
systolic dysfunction (Cardiac disorders) | 1 (1)
cardiomyopathy (Cardiac disorders) | 1 (1)
multiorgan failure (General disorders) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
Lung infection - pulmonary aspergillosis (Infections and infestations) | 1 (1)
skin infection - R leg cellulitis w/ abscess (Infections and infestations) | 1 (1)
Lung infection - Stenotrophomonas bacteremia (Infections and infestations) | 1 (1)
primary stenotrophomonas secondary AML (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No